CLINICAL TRIAL: NCT03763955
Title: Effectiveness of MIRT on Hand and Finger Dexterity in PD Patients
Acronym: H_F_ D_PD_MIRT
Status: Completed | Type: Observational
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Other Study IDs: H_F_D_PD_MIRT
Record Dates: First submitted 2018-11-26; First posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease; Dexterity; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PD patients: PD patients at 1-5 H&Y stage undergoes 4week Multidisciplinary Intensive Rehabilitation Treatment
  Interventions: Behavioral: MIRT

INTERVENTIONS:
Behavioral: MIRT — 4 week MIRT provide:
  1. front to front treatment (1 hour/day for 5 days/week)
  2. treatment with robotic devices (1 hour/day for 5 days/week)
  3. occupational therapy (1 hour/day for 5 days/week)
  Other Names: Multidisciplinary Intensive Rehabilitation Treatment

SUMMARY:
Aims of the study are (1) to evaluate the effectiveness of a specific OT treatment aimed to enhance finger and hand dexterity and (2) its impact on daily living autonomy of PD patients.

DETAILED DESCRIPTION:
Reduction in hand functionality and finger dexterity are significant, but often overlooked, symptoms of Parkinson's Disease (PD). They are strictly correlated with loss of patient's autonomy, due to their significant impact on Activities of Daily Living (ADL) and, consequently in patient's Quality of life (QoL). No studies investigated the effectiveness of a specific and functional-based Occupational Therapy (OT) treatment in improving hand functionality and finger dexterity in PD patients.

Aims of tthe study are to evaluate the effectiveness of a specific OT treatment aimed to enhance finger and hand dexterity and its impact on daily living autonomy of PD patients.

Retrospectively, 482 PD patients, hospitalized for a 4-week Multidisciplinary Intensive Rehabilitation Treatment (MIRT) between January 2015 and January 2018 were identified. All patients underwent 1h/day OT treatment. The outcome measure was the O'Connor finger dexterity test; secondary outcome measures were Minnesota dexterity test, UPDRS II and SPDDS scale. These measures were assessed at admission (T0) and discharge (T1).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's Disease

Exclusion Criteria:

* other neurological disease
* psychosis
* auditive or visual deficit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parkinsonian inpatients
Sampling Method: Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
O'Connor Finger Dexterity Test | 4 weeks
  peg-placement test aimed to evaluate the ability to manipulate small objects

SECONDARY OUTCOMES:
Minnesota Manual Dexterity Test | 4 weeks
  test aimed to evaluate the reach-to-grasp movements, gros manual dexterity and left vs right manual impairment